CLINICAL TRIAL: NCT06647953
Title: Prospective Treatment of Types I, II and III Pleuropulmonary Blastoma (PPB)
Brief Title: Testing a Standardized Approach to Surgery and Chemotherapy for Type I Pleuropulmonary Blastoma or the Addition of an Anti-cancer Drug, Topotecan, to the Usual Treatment for Types II and III Pleuropulmonary Blastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARAR2331; NCI-2024-08232 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARAR2331 (Other: Children's Oncology Group); ARAR2331 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Pleuropulmonary Blastoma
MeSH Terms: conditions — Pleuropulmonary blastoma | interventions — Specimen Handling; Cyclophosphamide; Dactinomycin; Dexrazoxane; Razoxane; Doxorubicin; Ifosfamide; Magnetic Resonance Spectroscopy; Watchful Waiting; Observation; Topotecan; High-Energy Shock Waves; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I, Arm 1 (VAC1200/VA regimen) (Experimental): Patients receive vincristine IV on days 1, 8, and 15 of cycles 1-3 and 5-7, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of each cycle, and cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1-4. Cycles repeat every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Tumor tissue is collected and centrally reviewed by a study pathologist. Patients also undergo blood sample collection, CT and ultrasound throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Procedure: Ultrasound Imaging; Drug: Vincristine
- Group I, Arm 2 (observation) (Active Comparator): Patients undergo observation on study. This includes tumor tissue collection and review by a study pathologist, and blood sample collection, chest CT, and ultrasound throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Patient Observation; Procedure: Ultrasound Imaging
- Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens) (Experimental): See Detailed Description for Group II, Arm 3.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Dexrazoxane; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Ifosfamide; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Topotecan; Drug: Vincristine
- Group II, Arm 4 (VTC400, IVADo, IVA regimens) (Experimental): See Detailed Description for Group II, Arm 4.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Dexrazoxane; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Ifosfamide; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Topotecan; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biospecimen Collection — Tumor tissue is collected and centrally reviewed by a study pathologist
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Group I, Arm 1 (VAC1200/VA regimen); Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
  Arms: Group I, Arm 1 (VAC1200/VA regimen); Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Drug: Dexrazoxane — Given IV
  Other Names: 2, 6-Piperazinedione, 4,4'-propylenedi-, (P)- (8CI); 2,6-Piperazinedione, 4, 4'-(1-methyl-1,2-ethanediyl)bis-, (S)- (9CI); ADR 529; ADR-529; ADR529; ICRF 187; ICRF-187; ICRF187; Razoxane (+)-form; Soluble ICRF (L-isomer)
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Group I, Arm 2 (observation)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
  Arms: Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
  Arms: Group I, Arm 1 (VAC1200/VA regimen); Group I, Arm 2 (observation)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Group I, Arm 1 (VAC1200/VA regimen); Group II, Arm 3 (VTC400, IVADo, VTC250, VAC1200 regimens); Group II, Arm 4 (VTC400, IVADo, IVA regimens)

SUMMARY:
This phase III trial tests how well surgery plus chemotherapy compared to surgery alone works in treating patients with type I pleuropulmonary blastoma (PPB), and tests how well surgery plus standard chemotherapy with the addition of topotecan works compared to surgery plus standard chemotherapy alone in treating patients with type II and III PPB.

Historically, most children with type I PPB had surgery and approximately 40% of children with type I PPB received chemotherapy following their surgery, usually for 22-42 weeks. There has not been a consistent standard for which children with type I PPB receive chemotherapy after surgery. For patients whose tumor has been removed completely with surgery, observation without chemotherapy may work as well as giving chemotherapy after surgery in preventing a return of the PPB tumor.

The standard chemotherapy for patients with types II or III PPB in the United States is four cycles of IVADo (ifosfamide, vincristine, dactinomycin, and doxorubicin) followed by 8 cycles of IVA (ifosfamide, vincristine and dactinomycin). Ifosfamide is in a class of medications called alkylating agents. It works by slowing or stopping the growth of tumor cells in the body. Vincristine is in a class of medications called vinca alkaloids. It works by stopping tumor cells from growing and dividing and may kill them. Dactinomycin is a type of antibiotic that is only used in cancer chemotherapy (antineoplastic antibiotic). It works by damaging the cell's deoxyribonucleic acid (DNA) and may kill tumor cells. Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's DNA and may kill tumor cells. It also blocks a certain enzyme needed for cell division and DNA repair. Topotecan is in a class of medications called topoisomerase I inhibitors. It works by interfering with tumor cell DNA which kills them. Giving topotecan in addition to standard IVADo and IVA chemotherapy regimens may shrink the cancer as well as or better than the standard therapy or could decrease the chance the tumor spreads while causing fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (complete response [CR] + partial response [PR]) to 2 cycles of window therapy with vincristine, topotecan and cyclophosphamide in children with Types II and III pleuropulmonary blastoma (PPB) using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

SECONDARY OBJECTIVES:

I. To estimate 3-year progression-free survival (PFS) and overall survival (OS) in children with Types II and III PPB.

II. To estimate 3-year PFS and OS in children with Type I PPB treated with surgery or surgery and chemotherapy using standardized guidelines.

EXPLORATORY OBJECTIVES:

I. To assess primary resection rate in children with Types I, II and III PPB using central radiology review and standardized surgical guidelines.

II. To assess surgical complications among those undergoing primary resection versus (vs.) biopsy followed by neoadjuvant chemotherapy for Types II and III PPB.

III. To establish a new cohort of prospectively treated children with newly diagnosed PPB which will serve as a comparison group for future novel agent trials.

IV. To evaluate toxicities in children treated for PPB including late cardiopulmonary toxicity.

V. To evaluate the molecular genetics/epigenetics of PPB and correlate with outcomes.

VI. To collect tumor tissue and serial blood samples for tumor profiling, liquid biopsies, and future correlative biology studies.

OUTLINE: Patients are assigned to 1 of 2 groups. For both groups, tumor tissue is centrally reviewed by a study pathologist. Blood samples are collected at specific clinical timepoints.

GROUP I (TYPE I/Ir PPB): Patients < 5 years old with Type I PPB whose tumor was not able to be completely removed by surgery are assigned to Arm 1. All other patients are assigned to Arm 2.

ARM 1 (VAC1200/VA REGIMEN): Patients receive vincristine intravenously (IV) on days 1, 8, and 15 of cycles 1-3 and 5-7, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of each cycle, and cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1-4. Cycles repeat every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, computed tomography (CT) and ultrasound throughout the study.

ARM 2: Patients undergo observation on study. This includes blood sample collection, chest CT, and ultrasound throughout the study.

GROUP II: (TYPE II/III PPB):

CYCLES 1-2 (VTC400 REGIMEN): Patients receive vincristine IV on days 1, 8, and 15 of each cycle, topotecan IV over 30 minutes on days 1-5 of each cycle, and cyclophosphamide IV over 15-30 minutes on days 1-5 of each cycle. Cycles repeat every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo multi-gated acquisition (MUGA) or echocardiography (ECHO), positron emission tomography (PET) or bone scan, CT, magnetic resonance imaging (MRI), and blood sample collection throughout the study.

Patients with complete response, partial response, or stable disease after cycle 2 are assigned to Arm 3. Patients with disease progression after cycle 2 are assigned to Arm 4. Patients also undergo surgery and radiation therapy as clinically indicated.

ARM 3:

CYCLES 3-6 (IVADo REGIMEN): Patients receive vincristine IV on day 1 of each cycle, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of each cycle, ifosfamide IV over 3 hours on days 1-2 of each cycle, dexrazoxane IV over 5-15 minutes on days 1-2 of each cycle, and doxorubicin IV over 3-15 minutes on days 1-2 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 7, 9, 11 (VTC250 REGIMEN): Patients receive vincristine IV on days 1, 8, and 15 of each cycle, topotecan IV over 30 minutes on days 1-5 of each cycle, and cyclophosphamide IV over 15-30 minutes on days 1-5 of each cycle. Treatment continues for 21 days every odd cycle for 3 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 8, 10, 12 (VAC1200 REGIMEN): Patients receive vincristine IV on day 1 of each cycle, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of each cycle, and cyclophosphamide IV over 30-60 minutes on day 1 of each cycle. Treatment continues for 21 days every even cycle for 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM 4:

CYCLES 3-6 (IVADo REGIMEN): Patients receive vincristine IV on day 1 of each cycle, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of each cycle, ifosfamide IV over 3 hours on days 1-2 of each cycle, dexrazoxane IV over 5-15 minutes on days 1-2 of each cycle, and doxorubicin IV over 3-15 minutes on days 1-2 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 7-12 (IVA REGIMEN): Patients receive vincristine IV on day 1 of each cycle, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of each cycle, and ifosfamide IV over 3 hours on day 1 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 24 months, then every 6 months until 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or younger
* Newly diagnosed PPB. Note that patients with known germline DICER1 variant or mosaicism with a large, solid unresectable thoracic mass with imaging features characteristic for Type II or III PPB are eligible without histologic confirmation of the diagnosis if a biopsy of the mass is not considered safe or feasible

  * Individuals are eligible based on institutional diagnosis of Type I, Ir, II or III PPB diagnosed within 60 days prior to enrollment. Children with Type II or III PPB at risk for clinical decompensation may receive protocol therapy while awaiting rapid central pathology review. Children with Type I or Ir PPB will be assigned to chemotherapy vs. observation based on imaging and central pathology review diagnosis. Type I and Ir patients should not begin chemotherapy prior to return of central pathology results
* For patients with Type II or III PPB (within 7 days prior to enrollment): A serum creatinine based on age/sex as follows:

  * Age: 1 month to < 6 months - Maximum Serum Creatinine (mg/dL): 0.4 (Male), 0.4 (Female)
  * Age: 6 months to < 1 year - Maximum Serum Creatinine (mg/dL): 0.5 (Male), 0.5 (Female)
  * Age: 1 to < 2 years - Maximum Serum Creatinine (mg/dL): 0.6 (Male), 0.6 (Female)
  * Age: 2 to < 6 years - Maximum Serum Creatinine (mg/dL): 0.8 (Male), 0.8 (Female)
  * Age: 6 to < 10 years - Maximum Serum Creatinine (mg/dL): 1 (Male), 1 (Female)
  * Age: 10 to < 13 years - Maximum Serum Creatinine (mg/dL): 1.2 (Male), 1.2 (Female)
  * Age: 13 to < 16 years - Maximum Serum Creatinine (mg/dL): 1.5 (Male), 1.4 (Female)
  * Age: ≥ 16 years - Maximum Serum Creatinine (mg/dL): 1.7 (Male), 1.4 (Female) OR - A 24 hour urine creatinine clearance ≥ 60 mL/min/1.73 m^2 OR - A glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)
  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* For patients with Type II or III PPB (within 7 days prior to enrollment): Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
* For patients with Type II or III PPB (within 7 days prior to enrollment): Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) ≤ 135 U/L

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Shortening fraction of ≥ 27% by echocardiogram, or ejection fraction of ≥ 50% by radionuclide angiogram (within 21 days prior to start of protocol therapy)
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible as long as they are NOT receiving anti-retroviral agents that are strong inhibitors or inducers of CYP3A4

Exclusion Criteria:

* Administration of prior PPB-directed chemotherapy is an exclusion criterion. Prior treatment for another malignancy is not an exclusion criterion
* Patients with known Charcot-Marie-Tooth disease
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response | Up to 2 cycles (cycles = 21 days) of window therapy with vincristine, topotecan and cyclophosphamide
  Response rates at the end of Cycle 2 will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method. Any eligible type II/III patients who do not undergo complete resection, have measurable disease at baseline (per central review) and start protocol therapy will be included in the primary analysis.

SECONDARY OUTCOMES:
Progression-free survival (PFS) in children with Types II and III pleuropulmonary blastoma (PPB) | From date of enrollment to the earliest occurrence of relapse, disease progression, or death due to any cause, assessed up to 3 years
  3-year PFS, along with the confidence intervals will be estimated using the Kaplan-Meier method. These results will be presented for Type II and III patients combined regardless of the timing of surgery.
Overall survival (OS) in children with Types II and III PPB | From date of enrollment to date of death due to any reason, assessed up to 3 years
  3-year OS, along with the confidence intervals will be estimated using the Kaplan-Meier method. These results will be presented for Type II and III patients combined regardless of the timing of surgery.
PFS in children with Types I PPB | From date of enrollment to the earliest occurrence of relapse, disease progression, or death due to any cause, assessed up to 3 years
  3-year PFS, along with the confidence intervals will be estimated using the Kaplan-Meier method.
OS in children with Types I PPB | From date of enrollment to date of death due to any reason, assessed up to 3 years
  3-year OS, along with the confidence intervals will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Resection rates for Type I PPB | Prior to protocol therapy
  Will be reported based on central radiology reviews.
Resection rates for Type II and III PPB | Prior to protocol therapy
  Will be reported based on central radiology reviews.
Resection rates for Type II and III PPB | Prior to cycle 5 (cycles = 21 days)
  Will be reported based on central radiology reviews.
Incidence of surgery-related adverse events | Up to 5 years
  Percentage of patients with surgery related adverse event. Results will be summarized separately for those undergoing primary resection versus those undergoing biopsy followed by neoadjuvant chemotherapy.
Incidence of adverse events | Up to 36 weeks
  Percentage of patients with Grade 3 or higher toxicities on protocol therapy.
PFS | Up to 5 years
  Will use Kaplan-Meier survival curves and log-rank tests to analyze PFS based on DICER1 germline status, hotspot mutations, and p53 status. Additionally, Cox proportional hazards regression will be used to evaluate the influence of these genetic factors on PFS controlling for confounding variables as necessary.
Primary outcome treatment effects by sex | Up to 5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% confidence intervals (CIs) by sex will be provided.
Primary outcome treatment effects by race | Up to 5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by race will be provided.
Primary outcome treatment effects by ethnicity | Up to 5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by ethnicity will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Ann P Schultz, Principal Investigator — Children's Oncology Group
Locations (72):
- United States (68):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Canada (4):
  - IWK Health Centre, Halifax, Nova Scotia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec